CLINICAL TRIAL: NCT01967212
Title: Swallowing Training Combined With Game-based Biofeedback in Post-stroke Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201210059RIC
Record Dates: First submitted 2013-10-13; First posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Dysphagia
Keywords: stroke; swallowing training; game-based; biofeedback
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Game-based swallow biofeedback (Experimental): swallowing training combined with game-based biofeedback in stroke dysphagia patient.
  Interventions: Device: Game-based swallow biofeedback
- Swallow training without biofeedback (Active Comparator)
  Interventions: Behavioral: Swallow training without biofeedback

INTERVENTIONS:
Device: Game-based swallow biofeedback — The intervention are divided into two parts：
  1. Traditional swallowing training 30 min by speech therapist.
  2. Game-based biofeedback combined with Mendelsohn's maneuver and effortful swallow 30 min by investigator.
  Other Names: The system was developed by Professor Chen, Jia-Jin and Dr. Li, Chih-Ming from Taiwan's National Cheng Kung University, Institute of Biomedical Engineering.
  Arms: Game-based swallow biofeedback
Behavioral: Swallow training without biofeedback — The intervention are divided into two parts：
  1. Traditional swallowing training 30 min by speech therapist.
  2. Mendelsohn's maneuver and effortful swallow without biofeedback 30 min.
  Arms: Swallow training without biofeedback

SUMMARY:
The purpose of this study is to determine whether swallowing training combined with game-based biofeedback is effective in the treatment of dysphagia due to stroke.

DETAILED DESCRIPTION:
Swallowing maneuvers are very effective if done correctly, but to evaluate the use of force and the extent of laryngeal elevation is very difficult.

The therapist often requests the patient to "swallow hard" or "maintain laryngeal elevation". However, it is difficult to provide appropriate feedback to the patient, because it's hard to see the throat muscle contraction and bone displacement,the real point of the force is not clear, only oral and tactile feedback is inadequate and when combined with sensory loss, fatigue or cognition impairment.

Biofeedback is defined as "the technique of using equipment (usually electronic) to reveal internal physiological events by visual and auditory signals, to teach patients to manipulate the intrinsic physiological activity (Basmajian, 1989).The rationale is thus that if a patient sees his muscle activity, rather than just feels his muscles contract, he will be able to contract his muscles more fiercely and therefore he will be able to train his muscles faster.

Past studies have shown that biofeedback can help nerve injury patients control their physiological activities such as swallowing training.

The purpose of this study is to determine whether swallowing training combined with game-based biofeedback is effective in the treatment of dysphagia due to stroke.

ELIGIBILITY:
Inclusion Criteria:

* stroke
* above 18 years-old
* pharyngeal stage dysphagia

Exclusion Criteria:

* on trachea
* cannot follow one command

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Hyoid bone displacement on the ultrasound | 6-8 weeks

SECONDARY OUTCOMES:
Swallow functional ability on the Functional Oral Intake Scale | 6-8 weeks

OTHER OUTCOMES:
SWAL-QOL Questionnaire | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tyng Guey Wang, PHD, Principal Investigator — Department of Physical Medicine and Rehabilitation,National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan